CLINICAL TRIAL: NCT00903149
Title: Long-term Effect of The Mother Infant Transaction Program (MITP)
Acronym: 2007/2/0150
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, Nina Margrethe Kynø, PhD, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Other Study IDs: 977468299
Record Dates: First submitted 2009-05-06; First posted 2009-05-18 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Premature Births
Keywords: Premature babies; Social interaction; Psychoeducative intervention; Mother Infant Transaction Program; Three years follow-up; Late preterm; Cognitive development; Social development; Emotional development; Motor development; Children born preterm and their parents
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MITP exposure or not: Mothers of children born preterm and term.

SUMMARY:
The purpose of this study is to investigate if a cost and time effective intervention in a previous RCT for preterm infants and their parents can reduce the parents experience of concern and stress, and improve the childrens development in various aspects at three years of corrected age.

Hypothesis 1: The preterm born children of parents who were enrolled in the earlier RCT have a higher developmental level then preterm children of parents who received the usual treatment.

Hypothesis 2: Parents who who were enrolled in the earlier RCT will have a lower level of stress and concern then parents who received treatment as usual.

DETAILED DESCRIPTION:
A previous RCT by Ravn (NCT00245843) investigated if the MITP could sensitize the mothers toward the babies signals and thereby increase the quality of joint attention. The study followed the children for 1 year.

This study is a follow-up to the above mentioned RCT. It investigates whether the effect of the RCT is present at three years corrected age.

The research questions are:

1. Can a psychoeducative program like the MITP influence the childrens' development in various aspects?
2. How did the MITP influence the parents experience of concern and stress three years later?
3. Were there any differences by the groups? a) Preterm intervention group b)Preterm control group c) Full term control group

The questionnaires to be used in this observational study are:

Ages and Stages

ELIGIBILITY:
Inclusion Criteria:

* All parents of children who participated in Ravn's RCT and who said yes to be asked for participation in an eventually later study will be asked.

Ages: 35 Months to 37 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The cohort is 42 preterm infants in the intervention group, 40 preterm and 40 full term in control groups.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Child development | 36 months
Parenting stress | Child age 36 months